CLINICAL TRIAL: NCT06829862
Title: Video-Guided Lifestyle Intervention Led by Patients' Own Doctor in Overweight and Obese Adult
Brief Title: Lifestyle Intervention on Patients With Overweight or Obesity
Acronym: LIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Profesor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-99
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Physical Activity; Eating Behavior; Therapeutic Alliance
MeSH Terms: conditions — Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Own Doctor Group (Experimental): The experimental group will receive access to audiovisual instructions (exercise and nutritional education) given by their specialist doctor.
  Interventions: Other: Own Doctor Education
- Unknown Doctor Group (Active Comparator): The control group will receive access to audiovisual instructions (exercise and nutritional education) given by an unknown doctor.
  Interventions: Other: Unknown Doctor Education

INTERVENTIONS:
Other: Own Doctor Education — The self-applied online program will comprise a 3-month behavioural intervention seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive access to the internet-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their specialist doctor.
  Arms: Own Doctor Group
Other: Unknown Doctor Education — The self-applied online program will comprise a 3-month behavioural intervention seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive the same intervention, but in this case supported by audiovisual instructions given by a doctor outside the patient.
  Arms: Unknown Doctor Group

SUMMARY:
This study aims to analyze the effects of a 3-month self-applied online program, focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on adults with obesity. Participants will be recruited by 8 doctors from 6 public Health Centers. These patients will be randomized allocated into two interventional groups: the experimental group will receive audiovisual instructions from their specialist doctor, and the control group from a doctor outside the patient. Assessment will include sociodemographic variables, body mass index, blood pressure, glycemic and lipid metabolism variables, physical activity level, adherence to the Mediterranean diet, therapeutic alliance, and health-related quality of life. The randomization process will be stratified according to BMI, therapeutic alliance, age, and sex.

DETAILED DESCRIPTION:
Obesity or being overweight, even other associated comorbidities, involve a worrying public health problem. The evidence shows that healthy eating and regular physical exercise, monitored by different means (internet, face to face, exercise diaries), play an important prevention role to maintain health while ageing. In this way, Information and Communication Technologies (ICTs) have been demonstrated as a useful tool to promote health, working on barriers at the same time, such as low motivation and difficulties maintaining regular exercise and/or healthy eating habits. ICTs also allows to reach a wider audience at a lower cost, due to their good cost-benefit relationship and the possibility of increasing the efficiency of interventions. Therefore, this study aims to analyze the effects of a 3-month self-applied online program, focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on adults with obesity. Participants will be recruited by 8 doctors from 6 public Health Centers. These patients will be randomized allocated into two interventional groups: the experimental group will receive audiovisual instructions from their specialist doctor, and the control group from a doctor outside the patient. Assessment will include sociodemographic variables, body mass index, blood pressure, glycemic and lipid metabolism variables, physical activity level, adherence to the Mediterranean diet, therapeutic alliance, and health-related quality of life. The randomization process will be stratified according to BMI, therapeutic alliance, age, and sex.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or grade I obesity (BMI > 25 and < 35).

Exclusion Criteria:

* No access to the Internet or a smartphone.
* Not having visited their doctor at least once in the last 2 years.
* Meeting DSM-IV-TR criteria for an Eating Disorder.
* Having a diagnosed serious psychological disorder (psychosis, bipolar disorder, major depressive disorder, substance abuse disorder, etc.).
* Having any disability that prevents or hinders exercise and physical activity.
* Receiving any weight loss treatment at another center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Body Mass Index (BMI) is a measure of body weight relative to height, calculated by dividing a person's weight in kilograms by the square of their height in meters.

SECONDARY OUTCOMES:
Blood Pressure | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Blood Pressure (BP) is the force exerted by circulating blood on the walls of the arteries. It is measured in millimeters of mercury (mmHg) and recorded as two values: systolic pressure (the pressure during heart contraction) over diastolic pressure (the pressure during heart relaxation).
Physical Activity Level | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Levels of Physical Activity will be assessed using the Short International Physical Activity Questionnaire (Short-IPAQ). This tool evaluates the frequency, duration, and intensity of physical activity, as well as sedentary behavior, in daily life. It estimates total physical activity in MET-min/week and records time spent sitting, providing a standardized measure of physical activity levels.
Adherence to the Mediterranean diet | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Adherence to the Mediterranean Diet will be assessed using the MEDAS (Mediterranean Diet Adherence Screener) from the PREDIMED study. This 14-item questionnaire evaluates adherence based on 12 questions about food consumption frequency and 2 questions on dietary habits associated with the Mediterranean diet. Each item is scored 0 or 1 point, with a total possible score ranging from 0 to 14 points. Higher scores indicate greater adherence.
Therapeutic Alliance | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Therapeutic Alliance will be assessed using the Working Alliance Inventory (WAI) questionnaire. This tool evaluates the relationship between a patient and their therapist across three key dimensions: (1) therapeutic goals, (2) tasks, and (3) therapeutic bond. Each item is scored on a Likert scale, with a total possible score ranging from low to high alliance strength. Higher scores indicate a stronger therapeutic alliance, which is associated with better treatment outcomes.
Health-related Quality of Life | Baseline (pre-intervention) and immediately post-intervention (3 months).
  Health-Related Quality of Life (HRQoL) will be assessed using the EuroQol-5D (EQ-5D) questionnaire. This tool evaluates five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on a multi-level scale. A health index score will be generated based on these dimensions. The visual analog scale (VAS) will not be used in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Fco. Lisón, Valencia, Valencia-valència, Spain